CLINICAL TRIAL: NCT01140165
Title: Effects of Hard Cheese and Butter on Markers of Cardiovascular Disease -A Randomized Controlled Dietary Human Intervention
Brief Title: Cheese and Human Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: The Danish Dairy Research Foundation, Denmark (Other); National Dairy Council (Other)
Responsible Party: Tine Tholstrup, Dpt Human Nutrition, University of Copenhagen, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A308
Record Dates: First submitted 2010-06-04; First posted 2010-06-09 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2009-10

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Cheese; Butter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- butter (Active Comparator): Danish butter
  Interventions: Other: cheese
- cheese (Experimental)
  Interventions: Other: cheese

INTERVENTIONS:
Other: cheese — the effect of cheese intake versus butter intake on blood lipids (primarily)
  Other Names: cheese, butter, dairy

SUMMARY:
The aim of this study is to examine if a diet rich in cheese will have a beneficial effect on risk markers of cardiovascular disease compared to a diet rich in butter.

The primary parameters are total cholesterol as well as LDL-, HDL cholesterol and triacylglycerol (TAG). The secondary parameters are hsCRP, markers of insulin resistance, fasting insulin and glucose (HOMA). Furthermore bloodpressure is measured.

ELIGIBILITY:
Inclusion Criteria:

* Sign written consent
* Age: 20-70
* BMI: 20-32
* Refrain from dietary supplements and blood donations prior to, and during the study

Exclusion Criteria:

* Known or suspected abuse of alcohol, drugs or medication
* Poor compliance
* Current or previously cardiovascular disease
* Diabetes Mellitus or other severe chronic disease, including severe allergies

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Total cholesterol | 6 weeks
LDL cholesterol | 6 weeks
HDL cholesterol | 6 weeks
Triglyceride | 6 weeks

SECONDARY OUTCOMES:
Insulin | 6 weeks
Glucose | 6 weeks
fasting hsCRP | 6 weeks
Blood pressure | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tine Tholstrup, PhD, Principal Investigator — Department of Human Nutrition, University of Copenhagen
Locations (1):
- Department of Human Nutrition, Frederiksberg, Denmark

REFERENCES:
- [Derived] Hjerpsted J, Leedo E, Tholstrup T. Cheese intake in large amounts lowers LDL-cholesterol concentrations compared with butter intake of equal fat content. Am J Clin Nutr. 2011 Dec;94(6):1479-84. doi: 10.3945/ajcn.111.022426. Epub 2011 Oct 26. PMID 22030228